CLINICAL TRIAL: NCT04969666
Title: A Phase II, Randomised, Double-Blind, Parallel-Group, Placebo-Controlled, Repeat Single Oral Dose Study of IPED2015 or Placebo in Otherwise Healthy Male Subjects With Erectile Dysfunction
Brief Title: A Phase II, Repeat Single Oral Dose Study of IPED2015 in Healthy Male Subjects With Erectile Dysfunction
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Initiator Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IPED2015CS02
Record Dates: First submitted 2021-06-28; First posted 2021-07-21 (Actual); Last update posted 2021-07-21 (Actual); Status verified 2021-06

CONDITIONS: Erectile Dysfunction
MeSH Terms: conditions — Erectile Dysfunction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- IPED2015_dose 1 (Experimental): Active treatment
  Interventions: Drug: IPED2015
- IPED2015_dose 2 (Experimental): Active treatment
  Interventions: Drug: IPED2015
- Placebo (Placebo Comparator): Placebo treatment
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: IPED2015 — Active treatment
  Arms: IPED2015_dose 1; IPED2015_dose 2
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This is a Phase II, randomised, double-blind, parallel-group, placebo-controlled study to investigate the effects of repeat single oral doses of IPED2015 in otherwise healthy male subjects with ED.

Up to 120 subjects are planned to be enrolled into 3 groups. Group 1 is planned to consist of 60 subjects, Group 2 is planned to consist of 36 subjects and Group 3 is planned to consist of 24 subjects. Groups 1, 2 and 3 will be conducted in parallel. Each subject will be dosed on four occasions. There will be three study treatments of dose 1 of IPED2015, dose 2 of IPED2015 or matched placebo. In each group, subjects will be randomised evenly to each of the three study treatments and will receive the same treatment on each visit.

DETAILED DESCRIPTION:
The primary objective of this study is to investigate the effects of repeat single oral doses of IPED2015 on male subjects with erectile dysfunction (ED) on ability to develop and maintain an erection.

ELIGIBILITY:
Inclusion Criteria:

Otherwise healthy male subjects with ED as determined from an IIEF-5 score of <16, with a body mass index of 18 to 35 kg/m2 (inclusive), of any ethnic origin.

Subject must have had at least one intent to have sexual intercourse during the last 3 months prior to Screening.

Exclusion Criteria:

Any significant CNS, cardiac, pulmonary, metabolic, renal, hepatic (including Gilbert's syndrome), gastrointestinal (GI) or psychiatric conditions, or history of fainting or syncope or such condition that, in the opinion of the Investigator, may place the subject at an unacceptable risk as a participant in the study, may interfere with the interpretation of safety or tolerability data obtained in this study, or may interfere with the absorption, distribution, metabolism or excretion of drugs, or with the completion of treatment according to this Protocol.

Clinically significant history of abnormal physical or mental health interfering with the study as determined by medical history and physical examinations obtained during Screening or Day -7 as judged by the Investigator (including [but not limited to], neurological, psychiatric, endocrine, cardiovascular, respiratory, GI, hepatic, or renal disorder).

Clinically significant abnormal laboratory results (including hepatic and renal panels, complete blood count, chemistry panel and urinalysis), 12-lead ECG and vital signs, or physical findings at Screening. In case of uncertain or questionable results, tests performed during the Screening visit may be repeated to confirm eligibility or judged to be clinically irrelevant for otherwise healthy subjects with ED.

Ages: 18 Years to 59 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-08-04 (Estimated); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-11-30 (Estimated)

PRIMARY OUTCOMES:
International Index of Erectile Function (IIEF-15) scale | 4 weeks
  Erectile Dysfunction assessment

SECONDARY OUTCOMES:
Rigiscan (diagnosis and assessment of male sexual impotence) | 4 weeks
  Device to assess erectile dysfunction
Semen analysis (check of quality of semen) | 4 weeks
  Analysis of tissue
Incidence of Treatment-Emergent Adverse Events | 4 weeks
  Assessment of patients health

CONTACTS AND LOCATIONS:
Overall Officials: Paul Westhead, MD, Principal Investigator — MAC UK

IPD SHARING:
Plan to Share IPD: No